CLINICAL TRIAL: NCT01976975
Title: Multi Level Analysis of Positive Valence Systems Across Mood Disorders
Brief Title: Brain Mechanisms of Human Motivation
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Diego A. Pizzagalli, Associate Professor, Department of Psychiatry, Harvard Medical School, Mclean Hospital
Other Study IDs: 2013-P-001352
Record Dates: First submitted 2013-10-25; First posted 2013-11-06 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Major Depressive Disorder; Bipolar Disorder
Keywords: Depression; Major Depressive Disorder; Bipolar Disorder; Mania; Hypomania; EEG; MRI; Reward
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression; Mania

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mood disorder patients: Patients with depressive and/or manic or hypomanic symptoms
- Healthy controls: Participants with no lifetime history of psychiatric illness

SUMMARY:
This study aims to investigate reward learning across the mood disorder spectrum and to investigate the predictive validity of reward learning for subsequent symptom severity.

DETAILED DESCRIPTION:
The study involves five sessions. In the first session, participants will play a computer task. In the second session, participants will go through a clinical interview and will have an EEG recording while playing another computer task. In the third session, participants will undergo an fMRI scan while playing another computer task. All tasks assess reward learning. At three and six months after the final session, participants will come back for a follow-up interview session during which a clinician will assess symptom severity. There will be no intervention in this study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Right-handed
* (For mood disorder group only) Stable medication over the past 8 weeks OR absence of any psychotropic medications for at least 2 weeks (for follow-up analyses testing effects in medication-free patients):

  * 6 weeks for fluoxetine,
  * 6 months for neuroleptics,
  * 2 weeks for benzodiazepines,
  * 2 weeks for any other antidepressants
  * 4 weeks for any mood-stabilizers

Exclusion Criteria:

* Suicidal ideation where outpatient treatment is determined unsafe by the study clinician
* Pregnant women or women of childbearing potential who 1) have not completed a negative urine pregnancy test prior to the MRI scan and/or 2) are seeking to become pregnant or believe that they may be pregnant
* Serious/unstable medical illness (e.g., cardiovascular, renal, endocrine, neurologic disease)
* Clinical or laboratory evidence of hypothyroidism
* History of seizure disorder, history or current diagnosis of dementia, score < 26 on the MMSE at screening
* History or current diagnosis of the following DSM-IV psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorder NOS, patients with mood congruent or mood incongruent psychotic features, anorexia nervosa, obsessive compulsive disorder
* Lifetime history of stimulant dependence (e.g., cocaine, amphetamines)
* Current use of Methylphenidate (Ritalin) and other ADHD medications with dopaminergic effects
* Patients with a lifetime history of electroconvulsive therapy (ECT)
* Failure to meet standard MRI safety requirements

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We are studying a population with depressive and/or manic or hypomanic symptoms, as well as healthy controls.
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2013-10; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diego A Pizzagalli, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pizzagalli D, Whitton A, Treadway M, Rutherford A, Kumar P, Ironside M, Kaiser R, Ren B, Dan R. Brain-based graph-theoretical predictive modeling to map the trajectory of transdiagnostic symptoms of anhedonia, impulsivity, and hypomania from the human functional connectome. Res Sq [Preprint]. 2023 Sep 28:rs.3.rs-3168186. doi: 10.21203/rs.3.rs-3168186/v1. PMID 37841877
- [Derived] Whitton AE, Kumar P, Treadway MT, Rutherford AV, Ironside ML, Foti D, Fitzmaurice G, Du F, Pizzagalli DA. Distinct profiles of anhedonia and reward processing and their prospective associations with quality of life among individuals with mood disorders. Mol Psychiatry. 2023 Dec;28(12):5272-5281. doi: 10.1038/s41380-023-02165-1. Epub 2023 Jul 4. PMID 37402852

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mood Disorder Patients | Healthy Controls
Started | 226 | 44
Completed | 79 | 32
Not Completed | 147 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mood Disorder Patients | Healthy Controls | Total
Number analyzed (Participants) | 226 | 44 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 3 | 11
  Between 18 and 65 years | 218 | 41 | 259
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 33 [18 to 64] | 30 [18 to 48] | 32 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 20 | 160
  Male | 86 | 24 | 110
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 22 | 11 | 33
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 32 | 4 | 36
  White | 144 | 27 | 171
  More than one race | 17 | 2 | 19
  Unknown or Not Reported | 9 | 0 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 226 | 44 | 270
Beck Depression Inventory-II [Mean (Full Range); unit: units on a scale] — Beck Depression Inventory-II (BDI-II). Measures the presence and severity of 21 depressive symptoms during the past two weeks, on a scale from 0 (none, or no change) to 3 (persistent, or worsening). Range: 0 to 63. Higher scores indicate greater symptom severity. Clinical categories for total score: 0-14: absent; 14-19: mild; 20-28: moderate; 29-63: severe.
  units on a scale | 27.87 [0 to 60] | .32 [0 to 4] | 22.59 [0 to 60]
Young Mania Rating Scale [Mean (Full Range); unit: units on a scale] — The YMRS is an 11-item scale that assesses manic symptoms based on the participant's report of his or her condition over the previous 48 hours, as well as the assessor's observations. The 11-items are elevated mood, increased motor activity-energy, sexual interest, sleep, irritability, rate/amount of speech, language-thought disorder, content, disruptive-aggressive behavior, appearance, and insight. The severity for 7-items are rated on a 5-point scale (0-4) and 4-items on a 9-point scale (0-8). The individual scores are summed for a total possible score of 0 (best) to 60 (worst). Population: The YMRS was not administered to subjects in the Healthy Control arm.
  units on a scale
    number analyzed (Participants) | 226 | 0 | 226
    (all) | 1.97 [0 to 22] |  | 1.97 [0 to 22]

OUTCOME MEASURES:

1. Primary Outcome: Change in Response Bias
Description: The Probabilistic Reward Task (PRT) is a behavioral task that measures an individual's ability to learn to choose a more rewarding outcome versus a less rewarding one (Response Bias). The response bias score is a ratio of the number of times a participant correctly chooses the high reward stimulus (the "rich" stimulus) versus the low reward stimulus (the "lean" stimulus). Response bias scores range between -1 and +1. A higher Response Bias score indicates a stronger bias toward the rich stimulus, and a negative Response Bias indicates a stronger bias toward the lean stimulus. The Change-in-Response-Bias is calculated by subtracting Response Bias in block 1 (trials 0-100) of the task from Response Bias in block 3 (trials 201-300) of the task. This metric represents the degree to which an individual is able to update behavior as a function of the asymmetrical reinforcement schedule.
Time Frame: Administered during the first session.
Population: Population includes patients and healthy controls who completed the PRT during the first session.
Measure: Mean (Full Range); unit: log-transformed ratio of scores
Arm/Group | Mood Disorder Patients | Healthy Controls
Number analyzed (Participants) | 135 | 34
log-transformed ratio of scores | .0546 [-.6194 to .7074] | .0787 [-.5408 to .7041]

2. Primary Outcome: Mean Accuracy on Gain Trials During an Instrumental Learning Task
Description: The instrumental learning task requires participants to choose between two abstract symbols. Each symbol in the pair is associated with an 80% or 20% probability of a given outcome (gain: win $1 or $0; loss: lose $1 or $0; neutral: view a gray square or see the word 'nothing'). The task consists of three blocks. Behavioral performance focuses on the number of times the participant chose the symbol that was associated more frequently associated with the more desirable outcome. A participant scores 1 if they choose correctly, and 0 if they choose in correctly, and correct choices across all three blocks are added and converted to a percentage relative to the total number of trials in that condition (i.e., gain, loss, or neutral). This study focused on percent of accuracy responses in the gain condition.
Time Frame: Administered in session 3 during 1.5 hour MR scan
Population: All participants who had readable Pessiglione task data
Measure: Mean (Full Range); unit: Percent of accurate responses
Arm/Group | Mood Disorder Patients | Healthy Controls
Number analyzed (Participants) | 77 | 31
Percent of accurate responses | 16.65 [10.33 to 21.33] | 17.03 [11.33 to 21.33]

3. Secondary Outcome: Symptom Severity at 6 Month Follow-up
Description: * Beck Depression Inventory (BDI-II). Severity of depressive symptoms, from 0 (no symptoms) to 63 (severely depressed)
  * Young Mania Rating Scale (YMRS). Severity of manic symptoms, from 0 (not manic) to 60 (severely manic)
  * Temporal Experience of Pleasure Scale (TEPS). The TEPS is an 18-item questionnaire. Ten items make up the TEPS-Anticipatory Pleasure scale with a range from 10 (not motivated) to 60 (highly motivated).
  * The other eight TEPS items make up the TEPS-Consummatory Pleasure scale; range from 8 (not responsive) to 48 (highly responsive)
  * Mood and Anxiety Symptom Questionnaire - Anhedonic Depression (MASQ-AD). The MASQ is a 62-item self-report on the severity of anxiety and depressive symptoms. The AD subscale is a 22-item measure of severity of anhedonic symptoms. Range: 22 -110 (higher scores mean greater severity)
  * Barrett Impulsiveness Scale 11 (BIS-11): a 30-item assessment of Trait Impulsivity. Range: 30-120 (higher scores mean more impulsiveness)
Time Frame: 6 months
Population: Population includes patients and controls who completed the 6-month follow up session
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Mood Disorder Patients | Healthy Controls
Number analyzed (Participants) | 68 | 30
units on a scale
  BDI-II | 15.24 [0 to 43] | .33 [0 to 4]
  YMRS | 1.41 [0 to 12] | .07 [0 to 1]
  TEPS Anticipatory Pleasure Scale | 39.41 [12 to 57] | 47.63 [38 to 58]
  TEPS Consummatory Pleasure Scale | 36.54 [8 to 48] | 40.30 [26 to 48]
  MASQ-AD; Anhedonic Depression severity | 70.59 [38 to 104] | 42.63 [22 to 69]
  BIS Impulsiveness | 67.47 [44 to 93] | 47.93 [38 to 59]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the date of subject consent until the conclusion of the 6-month follow-up interview (or until the subject was lost to contact).
Description: Definitions do not differ from the clinicaltrials.gov definition of adverse event.
Arm/Group | Mood Disorder Patients | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/226 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/226 | 0/44
Other Adverse Events (participants affected / at risk) | 0/226 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT01976975/Prot_SAP_000.pdf